CLINICAL TRIAL: NCT01759108
Title: Rebamipide for the Treatment of Xerostomia in Sjögren Syndrome
Brief Title: Rebamipide AND Sjögren Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, Principal investigator, University of Alexandria
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116619963
Record Dates: First submitted 2012-12-23; First posted 2013-01-02 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Improving Symptoms of Dry Mouth in Sjőgren's Syndrome
Keywords: xerostomia; rebamipide; efficacy; safety
MeSH Terms: conditions — Xerostomia | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rebamipide (Experimental): Patients will be randomized 1:1 to receive 300mg/d (100mg x3/day) of rebamipide for 12 weeks together with their usual therapy
  Interventions: Drug: Rebamipide
- Placebo (Placebo Comparator): Patients will be randomized 1:1 to receive 300mg/d (100mg x3/day) of placebo for 12 weeks together with their usual therapy.
  Interventions: Drug: Rebamipide

INTERVENTIONS:
Drug: Rebamipide — Patients will be randomized 1:1 to receive either 300mg/d (100mg x3/day) of rebamipide or placebo for 12 weeks together with their usual therapy.
  Other Names: Mucosta

SUMMARY:
Xerostomia is a major distressing symptom in Sjőgren's syndrome(SS). Preclinical and clinical studies have demonstrated an increase in saliva volume following rebamipide administration.We thus hypothesize that rebamipide may be efficacious in the treatment of dry mouth symptoms related to Sjőgren's syndrome.We will recruit SS patients in a randomized placebo-controlled trial for 12 weeks. The main outcome measure that will concern us is patient-assessed improvement of dry mouth symptoms and increase in salivary secretion Safety and efficacy was assessed at each visit.

DETAILED DESCRIPTION:
Xerostomia is a major distressing symptom in Sjőgren's syndrome (SS). Persistent dryness of the mouth causes oral pain, discomfort and significantly interferes with the quality of life. Rebamipide, in addition to its gastro-protective effect has displayed various anti-inflammatory actions including inhibition of neutrophilic leukocyte activation. Preclinical and clinical studies have demonstrated an increase in saliva volume following rebamipide administration.

The aim of the present study is to assess efficacy of rebamipide in the treatment of dry mouth symptoms related to Sjőgren's syndrome.

Methods: Fifty-five patients with American European Consensus Criteria Group (AECG)-based diagnosis of SS will participate in this randomized placebo-controlled trial. Inclusion criteria will include SS patients with dry mouth symptoms. Patients with dry mouth due to other conditions will be excluded. Patients will be randomized 1:1 to receive either 300mg/d (100mg x3/day) of rebamipide or placebo for 12 weeks together with their usual therapy. Outcome measures will include patient-assessed improvement of dry mouth symptoms and increase in salivary secretion (evaluation of unstimulated saliva; questionnaires including the visual analogue scale (VAS) for Sicca-syndrome VAS 0-100mm). Subjective and objective findings of dry mouth will be recorded at baseline, two, four, six, eight, ten and twelve weeks. Safety and efficacy will be assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* SS patients with dry mouth symptoms

Exclusion Criteria:

* Patients with dry mouth due to other conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
improvement of dry mouth symptoms | 12 weeks
  Improvement of dry mouth symptoms and increase in salivary secretion will be evaluated by questionnaires including the visual analogue scale (VAS) for Sicca-syndrome VAS 0-100mm.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abou-Raya, MD PhD, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt